CLINICAL TRIAL: NCT03122613
Title: A Double-blind, Randomized, Placebo-Controlled Trial of Curcumin Versus Placebo for Prevention of Relapse in Patients With Ulcerative Colitis
Brief Title: Curcumin for Prevention of Relapse in Patients With Ulcerative Colitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision made by team of investigators
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CUR2
Record Dates: First submitted 2017-04-07; First posted 2017-04-21 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Ulcerative Colitis in Remission
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinded using identical looking products in both arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curcumin (Active Comparator): Dietary supplements of Curcumin capsules
  Interventions: Dietary Supplement: Curcumin
- Curcumin Placebo (Placebo Comparator): Identical looking placebo of the active arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Curcumin — 3g of Curcumin per day
  Other Names: Turmeric
  Arms: Curcumin
Drug: Placebo — 3g of Curcumin Placebo per day
  Other Names: Curcumin placebo
  Arms: Curcumin Placebo

SUMMARY:
UC is a chronic inflammatory bowel disorder with relapsing and remitting course. The efficacy of mesalazine in preventing relapse in patients with UC is well-known and supported by randomized studies. However, mesalazine can be associated with side-effects. In addition, drug compliance is suboptimal, especially when disease is not active. Curcumin is a natural phytochemical derived from the Indian spice turmeric. It is widely used, has potent anti-inflammatory, anti-oxidant and anti-tumour properties.

The aims of this double-blind, placebo-controlled randomized trial is to assess the efficacy of curcumin in the prevention of relapse in patients with ulcerative colitis (UC).

DETAILED DESCRIPTION:
UC is a chronic inflammatory bowel disorder with relapsing and remitting course. The incidence of UC in Hong Kong has increased by 30-fold in the past three decades. The efficacy of mesalazine in preventing relapse in patients with UC is well-known and supported by randomized studies. However, mesalazine can be associated with side-effects. In addition, drug compliance is suboptimal, especially when disease is not active. Without mesalazine, the risk of relapse in UC in one year is approximately 60-70%. Repeated flares are disabling for the patient, and lead to increased hospitalisations, anatomical extension of disease, and increased cancer risk. In Hong Kong, 90 percent of patients with UC have low to medium compliance to mesalazine, and 50 percent would prefer the use of a complementary or alternative therapy to maintain disease remission. Identification of a natural product that is effective, acceptable, inexpensive and non-toxic remains an unmet need in patients with UC.

Curcumin is a natural phytochemical derived from the Indian spice turmeric. It is widely used, has potent anti-inflammatory, anti-oxidant and anti-tumour properties. Preclinical studies in experimental animals showed that curcumin is effective in preventing colitis. We reported in a randomized study that curcumin is effective in the induction of remission in patients with mild to moderately active UC. Although curcumin is popular amongst patients with inflammatory bowel disease, its efficacy in maintaining disease remission in UC is uncertain. We propose a double-blind, placebo-controlled trial to assess the efficacy of curcumin in preventing clinical relapse in patients with UC. Patients will be randomised to 2 gram curcumin once daily or an equivalent placebo for 12 months. The primary outcome is the rate of clinical relapse at 12 months. Secondary outcomes include adverse events, endoscopic remission, fecal calprotectin levels and time to relapse.

Because the use of curcumin is already popular in Asia, this important clinical question will not be a priority of pharmaceutical companies. If proven, this industry-independent trial will be a landmark study that identifies an alternative effective treatment to maintain disease remission in patients with UC. Regardless of the outcome, it will inform clinical practice and provide invaluable data to international guideline committees on the management of this chronic inflammatory disease.

The aims of this double-blind, placebo-controlled randomized trial is to assess the efficacy of curcumin in the prevention of relapse in patients with ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* in clinical remission for at least 1 month, defined as Mayo bowel frequency subscore ≤ 1 and Mayo rectal bleeding subscore = 0 (Table 2).
* a history of at least one flare with symptoms that required intervention within 24 months before screening
* age ≥ 18
* written informed consent obtained

Exclusion Criteria:

* receipt of immunosuppressive drugs or corticosteroids within 60 days of screening
* prior bowel surgery except appendectomy
* with severe relapse (Mayo score 9-12) in the last 3 months
* History or evidence of incompletely resected colonic mucosal dysplasia
* on regular curcumin supplements or intake of curry in diet for ≥5 days each week
* presence of infections (exclude simple infections such as influenza, etc.) or sepsis
* pregnancy or lactating women
* with a Mayo endoscopic subscore ≥2 on sigmoidoscopy or colonoscopy at baseline
* allergic to curry-related products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
The relapse rate at 12 months | 1 year
  Defined as clinical symptoms (increased bowel frequency with a bowel frequency Mayo subscore ≥ 1 or rectal bleeding with a Mayo rectal bleeding subscore ≥ 1) together with endoscopic evidence of active disease (Mayo endoscopic subscore ≥ 2).

SECONDARY OUTCOMES:
Adverse events | 1 year
  The severity grading of AEs will be assessed as Grade 1, 2, 3, 4 or 5 using the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 Grading Scale, which can be found at:
  http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE_4.03_2010-06-14_QuickReference_8.5x11.pdf
Endoscopic remission | 1 year
  Defined as a mayo endoscopic subscore of 0 or 1
Simple Clinical Colitis Activity Index (SCCAI) | 1 year
  compare the scores in two groups
Fecal calprotectin levels at 12 months | 1 year
  compare the difference of the levels between groups
Fecal immunochemical test (FIT) at 12 months | 1 year
  compare the positivity rate in those with flare
Quality of Life assessed by the Inflammatory Bowel Disease Questionnaire (IBDQ) | 1 year
  compare the scores in two groups
Patient Reported Outcomes (PRO) Questionnaire | 1 year
  The questionnaire will ask during the study follow up about the psychological aspects of UC patients, the baseline and score on final visit will be compared, as well as between the two groups
Pharmacokinetics study to measure the drug concentration-time courses | 1 year
  compare the absorption rate in two groups and to establish and evaluate the relationships and subsequently describe the effect-time courses of curcumin absorption in blood and colon.

CONTACTS AND LOCATIONS:
Overall Officials: Siew Ng, Prof., Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dignass A, Lindsay JO, Sturm A, Windsor A, Colombel JF, Allez M, D'Haens G, D'Hoore A, Mantzaris G, Novacek G, Oresland T, Reinisch W, Sans M, Stange E, Vermeire S, Travis S, Van Assche G. Second European evidence-based consensus on the diagnosis and management of ulcerative colitis part 2: current management. J Crohns Colitis. 2012 Dec;6(10):991-1030. doi: 10.1016/j.crohns.2012.09.002. Epub 2012 Oct 3. No abstract available. PMID 23040451
- [Background] Feagan BG, Macdonald JK. Oral 5-aminosalicylic acid for maintenance of remission in ulcerative colitis. Cochrane Database Syst Rev. 2012 Oct 17;10:CD000544. doi: 10.1002/14651858.CD000544.pub3. PMID 23076890
- [Background] Kane S, Huo D, Aikens J, Hanauer S. Medication nonadherence and the outcomes of patients with quiescent ulcerative colitis. Am J Med. 2003 Jan;114(1):39-43. doi: 10.1016/s0002-9343(02)01383-9. PMID 12543288
- [Background] Kane SV, Cohen RD, Aikens JE, Hanauer SB. Prevalence of nonadherence with maintenance mesalamine in quiescent ulcerative colitis. Am J Gastroenterol. 2001 Oct;96(10):2929-33. doi: 10.1111/j.1572-0241.2001.04683.x. PMID 11693328
- [Background] Sewitch MJ, Abrahamowicz M, Barkun A, Bitton A, Wild GE, Cohen A, Dobkin PL. Patient nonadherence to medication in inflammatory bowel disease. Am J Gastroenterol. 2003 Jul;98(7):1535-44. doi: 10.1111/j.1572-0241.2003.07522.x. PMID 12873575
- [Background] Leong RW, Lawrance IC, Ching JY, Cheung CM, Fung SS, Ho JN, Philpott J, Wallace AR, Sung JJ. Knowledge, quality of life, and use of complementary and alternative medicine and therapies in inflammatory bowel disease: a comparison of Chinese and Caucasian patients. Dig Dis Sci. 2004 Oct;49(10):1672-6. doi: 10.1023/b:ddas.0000043384.26092.f4. PMID 15573925
- [Background] Bernstein CN. Treatment of IBD: where we are and where we are going. Am J Gastroenterol. 2015 Jan;110(1):114-26. doi: 10.1038/ajg.2014.357. Epub 2014 Dec 9. PMID 25488896
- [Background] Hilsden RJ, Verhoef MJ, Rasmussen H, Porcino A, DeBruyn JC. Use of complementary and alternative medicine by patients with inflammatory bowel disease. Inflamm Bowel Dis. 2011 Feb;17(2):655-62. doi: 10.1002/ibd.21360. PMID 20848543
- [Background] Rawsthorne P, Clara I, Graff LA, Bernstein KI, Carr R, Walker JR, Ediger J, Rogala L, Miller N, Bernstein CN. The Manitoba Inflammatory Bowel Disease Cohort Study: a prospective longitudinal evaluation of the use of complementary and alternative medicine services and products. Gut. 2012 Apr;61(4):521-7. doi: 10.1136/gutjnl-2011-300219. Epub 2011 Aug 11. PMID 21836028
- [Background] Gupta SC, Kismali G, Aggarwal BB. Curcumin, a component of turmeric: from farm to pharmacy. Biofactors. 2013 Jan-Feb;39(1):2-13. doi: 10.1002/biof.1079. Epub 2013 Jan 22. PMID 23339055
- [Background] Vecchi Brumatti L, Marcuzzi A, Tricarico PM, Zanin V, Girardelli M, Bianco AM. Curcumin and inflammatory bowel disease: potential and limits of innovative treatments. Molecules. 2014 Dec 16;19(12):21127-53. doi: 10.3390/molecules191221127. PMID 25521115